CLINICAL TRIAL: NCT06992401
Title: An Observational Study Collecting Real-World Data on Intranasal IVIG Treatment in Long COVID-19 Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in Patients With Immunodeficiency Engaged in International Medical Tourism
Brief Title: Observational Study of Intranasal IVIG in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Patients Undergoing Medical Tourism
Acronym: IVIG-LC
Status: Not yet recruiting | Type: Observational
Sponsor: Tamara C Tamas (Other)
Responsible Party: Sponsor-Investigator, Tamara C Tamas, Director of Regulatory Affairs, Healing Hope International
Organization: Healing Hope International (Other)
Other Study IDs: HH-IVIG-LC001
Record Dates: First submitted 2025-05-23; First posted 2025-05-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Post-Acute Sequelae of SARS-CoV-2 Infection; Long COVID; Long COVID Fatigue; Long COVID Syndrome; COVID 19 Associated Coagulopathy; COVID-19 Vaccination
Keywords: Intranasal IVIG; Real-world data; Medical tourism; Long COVID fatigue; Cytokine panel; Immunoglobulin therapy; Brain fog; Chronic inflammation; Real-world evidence; Global health; Post-viral syndrome; Immune recovery
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mental Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long COVID Patients with Immunodeficiency: This group includes adult participants (ages 18-65) with a clinical diagnosis of Long COVID and laboratory-confirmed immunodeficiency (e.g., low IgG, low IgA, or specific antibody deficiency). Participants in this cohort are receiving intranasal immunoglobulin (IVIG) therapy as part of their standard care through international clinical sites. Data will be collected on treatment outcomes, cytokine and CRP profiles, antibody titers, and patient-reported symptoms including fatigue, cognitive function, and quality of life. No treatments are administered by the study team.

SUMMARY:
This observational study is being conducted by Healing Hope International to collect real-world data on an emerging treatment approach for Long COVID in patients with immunodeficiency. The study investigates the effects of intranasal immunoglobulin (IVIG) therapy in a real-world setting.

Participants will be individuals diagnosed with Long COVID who have confirmed immunodeficiency, such as low IgG or IgA levels or specific antibody deficiency. These individuals are receiving care through international clinical programs and will not receive any treatment as part of this study. Instead, Healing Hope will collect health information, clinical outcomes, and laboratory results from participating sites to better understand how intranasal IVIG might help reduce symptoms such as fatigue, brain fog, inflammation, and immune dysregulation.

The goal of this study is to contribute new insights into potential treatment options for Long COVID and to support responsible, science-backed care models for patients participating in medical tourism. No experimental drugs are being administered as part of this protocol. All treatment decisions are made independently by each clinical site. Data will be anonymized and used to advance knowledge in the field of immunological recovery and neuroinflammation.

DETAILED DESCRIPTION:
This observational study, initiated by Healing Hope International, is designed to collect real-world data (RWD) from individuals diagnosed with Long COVID who are undergoing clinical care involving intranasal immunoglobulin (IVIG) therapy at international medical tourism sites.

Eligible participants are adults (ages 18-65) with:

Persistent Long COVID symptoms for ≥12 weeks following SARS-CoV-2 infection,

Laboratory-confirmed immunodeficiency (e.g., low IgG/IgA, poor vaccine response, or specific antibody deficiency),

Elevated inflammatory biomarkers (e.g., CRP, cytokines),

No evidence of active infection (bacterial, viral, or fungal),

No comorbid neurological conditions (e.g., multiple sclerosis, Alzheimer's disease),

No current immunosuppressive therapies.

No investigational product will be administered by the study team. All treatments are prescribed and delivered independently by licensed international clinical sites. Healing Hope International operates as the sponsor and data coordinating center. Participants' data will be collected retrospectively and prospectively from site medical records, patient-reported surveys, and third-party laboratory assessments, including genetic testing for RXRA expression (e.g., via qPCR or NGS panels).

The primary data endpoints include:

Changes in immunological biomarkers (IgG/IgA, CRP, cytokine panel),

Clinical course of Long COVID symptoms (fatigue, cognitive impairment, respiratory issues),

Quality of life measures (collected via validated patient-reported outcome instruments).

The study complies with all applicable regulations for data protection and ethical research conduct, including informed consent, HIPAA-compliant data transfer where applicable, and de-identification of personal health information. Ethical approval will be obtained from an Institutional Review Board (IRB), and partner sites may obtain parallel local or national ethics approvals.

This study also seeks to characterize the broader landscape of medical tourism for regenerative therapies by mapping treatment accessibility, safety, and patient reported effectiveness in the context of international care. It does not replace or compete with regulated clinical trials but aims to generate actionable real world insights that can guide future controlled research.

By contributing to the body of evidence around global regenerative practices, this study supports the development of international ethical guidelines, compassionate use frameworks, and collaborative trial infrastructure in complex chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Clinical diagnosis of Long COVID (symptoms persisting ≥12 weeks after SARS-CoV-2 infection)
* Laboratory-confirmed immunodeficiency, including one or more of the following:
* Low serum IgG and/or IgA
* Specific antibody deficiency
* Low pneumonia titers
* Elevated inflammatory markers (e.g., CRP, cytokines)
* No active infections at the time of enrollment (bacterial, viral, or fungal)
* Negative for Lyme disease and NMDAR antibodies
* Willingness to provide informed consent for data collection and use

Exclusion Criteria:

* Current or recent active infection (e.g., viral, bacterial, or fungal)
* Use of immunosuppressive therapy within the last 3 months
* Active infections: Participants with active infections, including viral, bacterial, or fungal infections, will be excluded
* Neurological disorders: Participants with diagnosed neurological disorders (e.g., multiple sclerosis, Parkinson's disease, Alzheimer's disease) will be excluded
* Immunosuppressive therapy: Participants receiving immunosuppressive therapy will be excluded
* Inability to comply with study assessments or procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls adults aged 18 to 65 with persistent Long COVID symptoms and confirmed immunodeficiency, including low IgG/IgA or poor vaccine response. Participants must have elevated inflammatory markers and be free of active infections or neurological conditions. The population is observed while undergoing intranasal IVIG therapy internationally, with a focus on immunological, genetic, and quality of life outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue Severity Using the Fatigue Severity Scale (FSS) Using Patient-Reported Outcome Measures (PROMs) | Baseline and 12 Weeks
  Fatigue will be assessed using the Fatigue Severity Scale (FSS), a validated 9-item patient-reported outcome measure that evaluates the impact of fatigue on daily functioning. Each item is scored on a 7-point Likert scale. A decrease in total score from baseline indicates improvement.
Change in Cognitive Dysfunction Using the Cognitive Failures Questionnaire (CFQ) | Baseline and 12 Weeks
  Cognitive dysfunction (often referred to as "brain fog") will be evaluated using the Cognitive Failures Questionnaire (CFQ), a validated 25-item instrument that measures the frequency of cognitive lapses in daily activities. Higher scores indicate greater impairment. Improvement is reflected by a decrease in score.
Change in Breathlessness Using the Visual Analog Scale (VAS) | Baseline and 12 Weeks
  Breathlessness will be assessed using a Visual Analog Scale (VAS), in which participants rate their shortness of breath on a 100 mm line ranging from "no breathlessness" to "worst imaginable breathlessness." A lower score at 12 weeks compared to baseline indicates improvement.

SECONDARY OUTCOMES:
Change in C-Reactive Protein (CRP) Levels | Baseline and 12 Weeks
  Serum CRP levels will be collected at baseline and at 12 weeks to evaluate systemic inflammation. CRP is a sensitive marker of inflammatory activity. A reduction in CRP is considered a favorable outcome.
Change in Pro-Inflammatory Cytokines (e.g., IL-6, TNF-α, IL-1β) | Baseline and 12 Weeks
  Plasma cytokine levels will be analyzed at baseline and 12 weeks using multiplex assays. Changes in IL-6, TNF-α, and IL-1β will be assessed as indicators of neuroinflammation and systemic immune activation. Decreases suggest treatment benefit.
Change in Additional Cytokines and Inflammatory Markers | Baseline and 12 Weeks
  The following secondary cytokines and chemokines will also be tracked to evaluate the broader impact of intranasal IVIG on immune modulation. Reference ranges include:
  * Interferon-beta (IFN-β): <20.0 pg/mL
  * Interferon-gamma (IFN-γ): <60.0 pg/mL
  * Interferon-alpha (IFN-α): <20.0 pg/mL
  * Interleukin-10 (IL-10): <7.0 pg/mL
  * IL-18: ≤468 pg/mL
  * Monocyte Chemoattractant Protein-1 (MCP-1): ≤198 pg/mL
  * Macrophage Inflammatory Protein-1 alpha (MIP-1α): <220 pg/mL
  * Granulocyte-Monocyte Colony Stimulating Factor (GM-CSF): <15.0 pg/mL
  * IL-2 Receptor Alpha Soluble (sIL-2Rα): ≤959 pg/mL
  Changes in these markers will be analyzed to explore effects on neuroinflammatory signaling pathways, immune exhaustion, and cytokine resolution. Normalization trends will be documented and correlated with clinical improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anna Lara Kattan, MD: Regenerative Medicine, Principal Investigator — StemSolutions.mx

IPD SHARING:
Plan to Share IPD: Undecided
Healing Hope International is currently evaluating options for secure and ethical data sharing in accordance with international data protection standards and participant consent. If IPD sharing becomes feasible, de-identified data may be made available to qualified researchers upon request and IRB approval. A final determination will be made after assessing data governance infrastructure and stakeholder input.

REFERENCES:
- [Background] VanElzakker MB, Bues HF, Brusaferri L, Kim M, Saadi D, Ratai EM, Dougherty DD, Loggia ML. Neuroinflammation in post-acute sequelae of COVID-19 (PASC) as assessed by [11C]PBR28 PET correlates with vascular disease measures. Brain Behav Immun. 2024 Jul;119:713-723. doi: 10.1016/j.bbi.2024.04.015. Epub 2024 Apr 18. PMID 38642615
- [Background] Alaiya A, Alshukairi A, Shinwari Z, Al-Fares M, Alotaibi J, AlOmaim W, Alsharif I, Bakheet R, Alharbi L, Allam R, Asiri A, Memish Z, Alromaih K, Al-Mozaini M. Alterations in the Plasma Proteome Induced by SARS-CoV-2 and MERS-CoV Reveal Biomarkers for Disease Outcomes for COVID-19 Patients. J Inflamm Res. 2021 Sep 1;14:4313-4328. doi: 10.2147/JIR.S322430. eCollection 2021. PMID 34511970